CLINICAL TRIAL: NCT06759857
Title: A Randomized, Open, Positives Parallel-controlled, Multicenter Phase III to Evaluate the Efficacy and Safety of FHND9041 Versus Afatinib in First-line Treatment of Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: FHND9041 Versus Afatinib for Non-small Cell Lung Cancer
Acronym: FHND9041
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Chia Tai Fenghai Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FHND9041-III-01
Record Dates: First submitted 2024-12-23; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: FHND9041; phase Ⅲ
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FHND9041 (Experimental): Participants in this group will receive FHND9041, 80 mg orally, once daily, as first-line treatment for EGFR mutation-positive, locally advanced, or metastatic non-small cell lung cancer (NSCLC).
  Interventions: Drug: FHND9041
- Afatinib (Active Comparator): Participants in this group will receive afatinib, 40 mg orally, once daily, as first-line treatment for EGFR mutation-positive, locally advanced, or metastatic non-small cell lung cancer (NSCLC).
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: FHND9041 — FHND9041 is a novel therapeutic agent targeting EGFR mutations. Participants will take an 80 mg oral dose once daily until disease progression, intolerable toxicity, or meeting other study-defined discontinuation criteria.
  Arms: FHND9041
Drug: Afatinib — Afatinib is an approved, second-generation, irreversible EGFR tyrosine kinase inhibitor used as a standard first-line treatment for non-small cell lung cancer (NSCLC) with EGFR-sensitive mutations, such as L858R and Exon 19 deletions. Participants in this arm will take a 40 mg oral dose once daily. Afatinib serves as the active comparator in this study to evaluate the efficacy and safety of FHND9041.
  Arms: Afatinib

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness and safety of FHND9041 compared to afatinib as first-line treatments for epidermal growth factor receptor mutation-positive (EGFRm+) locally advanced or metastatic non-small cell lung cancer (NSCLC). The main questions it aims to answer are:

* Does FHND9041 improve progression-free survival (PFS) compared to afatinib?
* Are there differences in safety profiles between FHND9041 and afatinib?

Researchers will compare FHND9041 (80 mg, orally, once daily) with afatinib (40 mg, orally, once daily) in a randomized, open-label, parallel-controlled, multicenter Phase III trial.

Participants who meet the inclusion criteria, including having EGFR mutations (L858R and/or Exon 19 deletion) and no prior treatment, will be randomly assigned in a 1:1 ratio to either the FHND9041 group or the afatinib group. Treatment will continue until disease progression, intolerable drug-related toxicity, or other pre-specified treatment discontinuation criteria are met.

Study Procedures:

Participants will:

* Be screened for eligibility and randomly assigned to one of two groups.
* Receive study drugs per their assigned group.
* Undergo regular tumor assessments by Response Evaluation Criteria in Solid Tumors, version 1.1( RECIST 1.1) every six weeks during the first 18 cycles, then every nine weeks until disease progression. For intracranial efficacy, Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM ) criteria will be applied.
* Participate in pharmacokinetic studies (FHND9041 group only) with blood samples collected pre-dose at specified cycles and on the day of discontinuation.

After disease progression, participants will be followed for survival every three months.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥ 18 years, with no gender restrictions.
* Histologically or cytologically confirmed diagnosis of locally advanced or metastatic non-small cell lung cancer (NSCLC), including patients with recurrent disease following prior surgical treatment or newly diagnosed Stage IIIb, IIIc, or IV NSCLC (staging based on the 8th edition of the AJCC guidelines).
* No prior systemic anti-tumor therapy (e.g., standard chemotherapy, targeted therapy, biological therapy, or immunotherapy). Patients who have received adjuvant or neoadjuvant therapy (chemotherapy, radiotherapy, or other treatments) are eligible if disease progression occurred at least 6 months after completing the prior treatment.
* Presence of a confirmed EGFR-positive gene mutation sensitive to EGFR-TKI treatment, including exon 19 deletion or L858R mutation.
* At least one measurable tumor lesion at baseline that meets the following criteria:

No prior radiotherapy or biopsy during the screening period (if the subject has only one measurable lesion, fine-needle aspiration cytology to confirm genetic status is permitted; however, baseline imaging must be performed at least 7 days after the biopsy).

Lesion can be accurately measured with a longest diameter ≥ 10 mm (or a short axis ≥ 15 mm for lymph nodes).

Lesion can be assessed using CT or MRI, with the same imaging modality used consistently for subsequent evaluations.

* An Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
* A life expectancy of ≥ 3 months.
* Female participants of childbearing potential must have a negative serum pregnancy test prior to enrollment. Male and female participants with reproductive potential must agree to maintain abstinence or use effective contraception during the study and for at least 3 months following the last dose of the investigational drug.
* Participants must demonstrate the ability to understand the study objectives and procedures, comply with protocol requirements, cooperate with study-related visits, and provide written informed consent, indicating their voluntary participation.

Exclusion Criteria:

● Pre-treatment History: Major Surgery: Subjects who have undergone major surgery within 28 days before the first dose of the study drug. For the purposes of this study, major surgery refers to level 3 and level 4 surgeries as defined in the "Administrative Measures for the Clinical Application of Medical Technology" (implemented on May 1, 2009).

Radiotherapy: Subjects who have received local radiotherapy or palliative radiotherapy for bone metastasis within 14 days prior to the first dose of the study drug.

CYP3A4 Interactions: Subjects who have received a strong CYP3A4 inhibitor or a strong inducer within 7 days before the first dose, or who need to continue using these drugs during the study period.

Chinese Herbal Medicines: Subjects who have received Chinese herbal medicines or proprietary Chinese medicine preparations for anti-tumor indications within 7 days prior to the first dose, or who need to continue using these during the study period.

QT Prolongation Medications: Subjects who are receiving drug treatments known to prolong the QTc interval or potentially cause torsades de pointes, and who need to continue using these medications during the study period.

* Unhealed Toxicity: Subjects who have unresolved toxic reactions of grade ≥ 2 (according to NCI-CTCAE 5.0 standards) related to previous treatments, except for hair loss and grade 2 neuropathy caused by platinum-based drugs.
* Spinal Cord Compression/Brain Metastases:

Subjects with spinal cord compression or brain metastases, except those who are asymptomatic, stable, and have not required steroid treatment for at least 4 weeks prior to the start of the study.

Subjects with brain metastases who have received local radiotherapy must show stable symptoms for at least 28 days following completion of the radiotherapy.

* Uncontrolled Systemic Diseases: Subjects with severe or uncontrolled systemic diseases (e.g., hypertension not controlled by medication, active bleeding disorders) that, in the investigator's opinion, may interfere with the participant's ability to comply with the study protocol.
* Active Infections:

Subjects with active infections that require medical treatment, including HBV (HBsAg positive, HBV-DNA > 1000 cps/ml or 200 IU/ml, and AST or ALT > 2.0 ULN), HCV (HCV antibody positive and HCV-RNA ≥ 1000 IU/mL), HIV, syphilis, or other serious infections.

● Gastrointestinal Dysfunction: Subjects with clinically significant gastrointestinal issues that may affect the intake, transport, or absorption of the study drug. This includes inability to take oral medication, uncontrolled nausea or vomiting, history of extensive gastrointestinal resection, unresolved recurrent diarrhea, or gastrointestinal diseases such as Crohn's disease or ulcerative colitis requiring long-term use of proton pump inhibitors (PPI).

● Cardiac Exclusion Criteria: QTc Prolongation: Subjects with an average QT interval (QTcF) corrected by Fridericia's formula greater than: 450 ms for males; 470 ms for femaleS; ECG Abnormalities: Subjects with clinically significant arrhythmias, heart block, or other abnormalities in resting ECG, such as complete left bundle branch block, third-degree heart block, second-degree type II block, PR interval > 250 ms, or recent myocardial infarction within 6 months; Risk Factors for QTc Prolongation: Subjects with factors increasing the risk of QTc prolongation or arrhythmia, such as heart failure, moderate or severe hypokalemia, congenital long QT syndrome, family history of sudden cardiac death under 40 years of age, or concurrent use of drugs that may prolong the QT interval; Left Ventricular Ejection Fraction (LVEF) ≤ 50%.

* Interstitial Lung Disease (ILD): History of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis requiring steroid treatment, or clinically active ILD.
* Bone Marrow or Organ Dysfunction:Subjects who do not meet the laboratory standards for organ function, including but not limited to: Neutrophil count < 1.5 x 10^9/L; Platelet count < 90 x 10^9/L; Hemoglobin < 90 g/L;ALT or AST > 2.5 times the upper limit of normal (ULN), or > 5 times ULN in cases of liver metastasis ;Serum total bilirubin > 1.5 times ULN (or > 3 times ULN if the subject has Gilbert syndrome or liver metastasis); Creatinine > 1.5 times ULN, with a creatinine clearance rate < 50 mL/min (confirmed by Cockcroft-Gault formula, if creatinine is > 1.5 times ULN).
* Allergic Reactions: Subjects with a known history of allergy or hypersensitivity to the active ingredients or excipients of the study drug, or to drugs with similar chemical structures to the investigational drug.
* Lactating Women: Lactating women are excluded from participation.
* Other Malignant Tumors: Subjects with a history of other malignant tumors, except for those with clinically cured cervical carcinoma in situ, basal cell carcinoma, squamous cell skin cancer, or papillary thyroid carcinoma within the past 5 years.
* Serious Eye Diseases: Subjects with any serious or uncontrolled eye disease that may increase the safety risk of the investigational drug, as determined by the investigator.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-03-04 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 24 months
  The time from randomization to the first documented disease progression ( assessed by investigators) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  The proportion of participants with confirmed complete response (CR) or partial response (PR)
Overall Survival (OS) | 36 months
  The time from randomization to death due to any cause.
Duration of Response (DoR) | 24 months
  The time from the first documented CR or PR to the first documented disease progression or death, whichever occurs first.
Disease Control Rate (DCR) | 24 months
  The proportion of participants with confirmed CR, PR, or stable disease (SD) for at least 6 weeks
Depth of Response (DepOR) | 24 months
  The maximum percentage change in the sum of target lesion diameters from baseline
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 ( EQRTC-C30) | 24 months
  Change from baseline in quality of life (QoL) scores using the EQRTC-C30 questionnaire. The scale ranges from 0 to 100, where higher scores indicate better quality of life.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Lung Cancer Module 13(LC13) | 36 months
  Change from baseline in quality of life (QoL) scores using the LC13 questionnaire. The scale ranges from 0 to 100, where higher scores indicate better quality of life.
Lung Cancer Symptom Scale(LCSS) | 36 months
  Change from baseline in quality of life (QoL) scores using the LCSS questionnaire. The scale ranges from 0 to 100, where higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Soria JC, Felip E, Cobo M, Lu S, Syrigos K, Lee KH, Goker E, Georgoulias V, Li W, Isla D, Guclu SZ, Morabito A, Min YJ, Ardizzoni A, Gadgeel SM, Wang B, Chand VK, Goss GD; LUX-Lung 8 Investigators. Afatinib versus erlotinib as second-line treatment of patients with advanced squamous cell carcinoma of the lung (LUX-Lung 8): an open-label randomised controlled phase 3 trial. Lancet Oncol. 2015 Aug;16(8):897-907. doi: 10.1016/S1470-2045(15)00006-6. Epub 2015 Jul 5. PMID 26156651
- [Background] Schuler M, Paz-Ares L, Sequist LV, Hirsh V, Lee KH, Wu YL, Lu S, Zhou C, Feng J, Ellis SH, Samuelsen CH, Tang W, Marten A, Ehrnrooth E, Park K, Yang JC. First-line afatinib for advanced EGFRm+ NSCLC: Analysis of long-term responders in the LUX-Lung 3, 6, and 7 trials. Lung Cancer. 2019 Jul;133:10-19. doi: 10.1016/j.lungcan.2019.04.006. Epub 2019 Apr 8. PMID 31200814
- [Background] Guo Y, Ahn MJ, Chan A, Wang CH, Kang JH, Kim SB, Bello M, Arora RS, Zhang Q, He X, Li P, Dechaphunkul A, Kumar V, Kamble K, Li W, Kandil A, Cohen EEW, Geng Y, Zografos E, Tang PZ. Afatinib versus methotrexate as second-line treatment in Asian patients with recurrent or metastatic squamous cell carcinoma of the head and neck progressing on or after platinum-based therapy (LUX-Head & Neck 3): an open-label, randomised phase III trial. Ann Oncol. 2019 Nov 1;30(11):1831-1839. doi: 10.1093/annonc/mdz388. PMID 31501887
- [Background] Paz-Ares L, Tan EH, O'Byrne K, Zhang L, Hirsh V, Boyer M, Yang JC, Mok T, Lee KH, Lu S, Shi Y, Lee DH, Laskin J, Kim DW, Laurie SA, Kolbeck K, Fan J, Dodd N, Marten A, Park K. Afatinib versus gefitinib in patients with EGFR mutation-positive advanced non-small-cell lung cancer: overall survival data from the phase IIb LUX-Lung 7 trial. Ann Oncol. 2017 Feb 1;28(2):270-277. doi: 10.1093/annonc/mdw611. PMID 28426106
- [Background] Schuler M, Yang JC, Park K, Kim JH, Bennouna J, Chen YM, Chouaid C, De Marinis F, Feng JF, Grossi F, Kim DW, Liu X, Lu S, Strausz J, Vinnyk Y, Wiewrodt R, Zhou C, Wang B, Chand VK, Planchard D; LUX-Lung 5 Investigators. Afatinib beyond progression in patients with non-small-cell lung cancer following chemotherapy, erlotinib/gefitinib and afatinib: phase III randomized LUX-Lung 5 trial. Ann Oncol. 2016 Mar;27(3):417-23. doi: 10.1093/annonc/mdv597. Epub 2015 Dec 8. PMID 26646759
- [Background] Sequist LV, Yang JC, Yamamoto N, O'Byrne K, Hirsh V, Mok T, Geater SL, Orlov S, Tsai CM, Boyer M, Su WC, Bennouna J, Kato T, Gorbunova V, Lee KH, Shah R, Massey D, Zazulina V, Shahidi M, Schuler M. Phase III Study of Afatinib or Cisplatin Plus Pemetrexed in Patients With Metastatic Lung Adenocarcinoma With EGFR Mutations. J Clin Oncol. 2023 Jun 1;41(16):2869-2876. doi: 10.1200/JCO.22.02547. PMID 37235976
- [Background] Harvey RD, Adams VR, Beardslee T, Medina P. Afatinib for the treatment of EGFR mutation-positive NSCLC: A review of clinical findings. J Oncol Pharm Pract. 2020 Sep;26(6):1461-1474. doi: 10.1177/1078155220931926. Epub 2020 Jun 20. PMID 32567494